CLINICAL TRIAL: NCT00712595
Title: Mifepristone 5 mg Versus 10 mg for the Treatment of Uterine Leiomyomata. A Randomized, Double Blinded Clinical Trial.
Brief Title: Mifepristone for Treatment of Uterine Fibroids
Acronym: Mifemyo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mediterranea Medica S. L. (Other)
Responsible Party: Dr. Josep Lluis Carbonell i Esteve, Mediterranea Medica S. L.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mife_Fibroids_01
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; mifepristone; antiprogestins
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mifepristone 10 mg daily for three months
  Interventions: Drug: Mifepristone
- 2 (Experimental): Mifepristone 5 mg daily for three months
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Oral administration of Mifepristone 10 mg daily for three months
  Other Names: Low doses of antiprogestins to treat uterine fibroids.
  Arms: 1
Drug: Mifepristone — Oral administration of Mifepristone 5 mg, daily for three months
  Arms: 2

SUMMARY:
The objectives of this study are to estimate the efficacy and safety of the daily administration of mifepristone 5 mg versus 10 mg for three months for the treatment of uterine fibroids.

The hypothesis of the study is that both mifepristone doses reduce the volume of the myoma in about 40% after 3 months of treatment.

DETAILED DESCRIPTION:
Women, in fertile age or in premenopausal status, presenting symptomatic uterine fibroids were randomly assigned to receive 5 mg or 10 of mifepristone.

The diminishing of prevalence of symptoms attributable to uterine fibroids is the most important goal to achieve under both treatments. The possible side effects of mifepristone are slight and women's adherence to treatment is remarkable. Also the reduction of the volumes of the uterus and fibroids contribute to enhance the wellbeing of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine leiomyomata
* Reproductive age or premenopausal
* Accepting the use of non hormonal contraception
* Conformity in keeping a monthly log of all episodes of vaginal bleeding during the treatment as well as all side effects of mifepristone
* Agreeing to have ultrasound examinations in every follow-up or evaluation visit
* Agreeing to two endometrial biopsies: one before starting treatment and another in the following 10 days after treatment termination.

Exclusion Criteria:

* Pregnancy or desire to become pregnant
* Breastfeeding
* Hormonal contraception or any hormonal therapy received in the last three months
* Signs or symptoms of pelvic inflammatory disease
* Adnexal masses
* Abnormal or unexplained vaginal bleeding
* Suspected or diagnosed malignant neoplastic disease
* Signs or symptoms of mental illness
* Adrenal disease
* Sickle cell anemia
* Hepatic disease
* Renal disease
* Coagulopathy
* Any other severe or important disease
* Any contraindication to receiving antiprogestins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Volume of the uterine leiomyomata with 5 mg versus 10 mg daily of mifepristone after 3 months of treatment | 3 months

SECONDARY OUTCOMES:
Volume of the uterus with 5 mg versus 10 mg daily of mifepristone after 3 months of treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep LL. Carbonell, MD, Principal Investigator — Mediterranea Medica
Locations (1):
- Hospital Eusebio Hernández, Havana, Ciudad Habana, Cuba